CLINICAL TRIAL: NCT04159441
Title: Hepatotoxicity of Antituberculosis Therapy in a Real-World Setting: an Observational Study in China
Brief Title: Hepatotoxicity of Antituberculosis Therapy (HAT) Study
Acronym: HAT
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Huashan Hospital (Other)
Responsible Party: Principal Investigator, Wen-hong Zhang, Director of Division of Infectious Diseases, Huashan Hospital
Other Study IDs: RWD-017
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2019-11-12 (Actual); Status verified 2019-11

CONDITIONS: Chemical and Drug Induced Liver Injury
Keywords: Hepatotoxicity of Antituberculosis Therapy; DILI
MeSH Terms: conditions — Chemical and Drug Induced Liver Injury

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Biospecimen Retention: None Retained — Blood
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Other: None intervetion — None intervetion

SUMMARY:
Drug-induced liver injury (DILI) is a common side effect in antituberculosis therapy, which interuputs the treatment of TB and leads to a higher proportion of Multidrug-Resistence TB(MDR-TB).The study primalily aims to observe the proportion of DILI in antituberculosis therapy. Furthermore, the secondary objective is to study the proportion of liver injury of based liver disase,liver failure and adjustment of chemotherapy in the obersevational study.

DETAILED DESCRIPTION:
Drug-induced liver injury (DILI) is a common side effect in antituberculosis therapy, which interuputs the treatment of TB and leads to a higher proportion of Multidrug-Resistence TB(MDR-TB).The study primalily aims to observe the proportion of DILI in antituberculosis therapy. Furthermore, the secondary objective is to study the proportion of liver injury of based liver disase,liver failure and adjustment of chemotherapy in the obersevational study.

ELIGIBILITY:
Inclusion Criteria:

* 1) Patients who are about to start anti-tuberculosis treatment 2) Male or female, age > 18 years old 3) Voluntary signing of "Subject Informed Consent Form"

Exclusion Criteria:

- 1)A history of taking anti-tuberculosis drugs within 6 months before the treatment; 2)Abnormal liver function before starting anti-tuberculosis treatment; 3)DILI at the time of enrollment. 4)Combined with malignant tumors (including hematological tumors), HIV infection, etc.

5) According to the investigator's judgment, patients who cannot complete this study or who cannot comply with the requirements of this study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who are about to start anti-tuberculosis treatment in the real world, including combined with different kinds of based disease, such as viral hepatitis,systematic infection,etc.
Sampling Method: Probability Sample
Enrollment: 5000 (Estimated)
Dates: Start 2019-12-05 (Estimated); Primary Completion 2020-12-05 (Estimated); Study Completion 2021-06-05 (Estimated)

PRIMARY OUTCOMES:
Proportion of DILI in antituberculosis therapy | 12 months(DILI occurs) or 24 months(None-DILI occur) after treatment initiation
  The study primalily aims to observe the proportion of DILI in antituberculosis therapy,by monitoring and following up the liver function of the participants.

SECONDARY OUTCOMES:
Proportion of liver injury of based liver disase,liver failure and adjustment of chemotherapy | 12 months(DILI occurs) or 24 months(None-DILI occur) after treatment initiation
  The study secondly aims to observe the proportion of liver injury of based liver disase,liver failure and adjustment of chemotherapy,by monitoring and following up the liver function, drug treatment of the participants.

CONTACTS AND LOCATIONS:
Overall Officials: Wenhong Zhang, Study Chair — Huashan Hospital; Yongguo LI, Principal Investigator — First Affiliated Hospital of Harbin Medical University; Dapeng Bai, Principal Investigator — Haihe Hospital in Tianjin; Meiying Wu, Principal Investigator — The Fifth Hospital in Suzhou; Huaicheng Wang, Principal Investigator — Third People's Hospital in Changzhou; Qinfang Ou, Principal Investigator — Fifth Hospital in Wuxi; Yonglan Pu, Principal Investigator — First People's Hospital in Taicang; Fan Xia, Principal Investigator — The 905th Hospital of the PLA Navy; Yuanyuan Chen, Principal Investigator — Red Cross Hospital, Hangzhou, China; Zumo Zhou, Principal Investigator — People's Hospital in Zhuji; Xiaohong Chen, Principal Investigator — Fuzhou Pulmonary Hospital in Fujian; Guofang Deng, Principal Investigator — The Third People's Hospital in Shenzhen; Shiwu Ma, Principal Investigator — People's Liberation Army Joint Service Support Unit 920 Hospital (formerly Kunming General Hospital of Chengdu Military Region); Youfang Gao, Principal Investigator — People's Hospital in Haozhou; Yongfang Jiang, Principal Investigator — Central South University Xiangya Second Hospital; Hongying Yu, Principal Investigator — Huaihua First People Hospital in Hunan; Bo Chen, Principal Investigator — Longtan Hospital in Guangxi; Weiqiang Zheng, Principal Investigator — Guangdong Medical University Affiliated Hospital; Liyuan Zhang, Principal Investigator — The Second Affiliated Hospital of Hainan Medical College; Guanghui Xu, Principal Investigator — Tuberculosis Control Center in Jiangmen; Anjie Zhang, Principal Investigator — Yubei Second People's Hospital; Hancheng Liang, Principal Investigator — The Sixth People's Hospital in Dongguan; Yuqing Wu, Principal Investigator — Chest Hospital in Jiangxi; Xilin Zhang, Principal Investigator — The Forth People's Hospital in Foshan

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: CSR